CLINICAL TRIAL: NCT03526068
Title: The First in the World Human Proof-of-concept Study on Disinfection and Healing Acceleration Capabilities of 222nm Wave Length Narrow Band Ultraviolet Lighting Device
Brief Title: Proof-of-concept Study on Disinfection and Healing Acceleration Capabilities of 222nm Wave Length Narrow Band Ultraviolet Lighting Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: USHIO. INC (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/00105-AMD0001
Record Dates: First submitted 2018-04-17; First posted 2018-05-16 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-04

CONDITIONS: Ultraviolet Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SafeZoneUVC (Experimental): Patients were subjected to 90s UV light therapy of 540 mW/cm2 sessions 2 times a week for 2 weeks for a total of 4 sessions. Pre and post UV light therapy swabs were taken after standard wound irrigation
  Interventions: Device: SafeZoneUVC

INTERVENTIONS:
Device: SafeZoneUVC — SafeZoneUVC® uses a Krypton Chloride (Kr-Cl) excimer lamp as its light source. The Kr-Cl excimer lamp emits UVC light having a main wavelength of 222 nm when the Kr-Cl exciplex is deactivated to non-excited state molecule in the lamp. This 222 nm UVC light can inactivate bacteria, while the Kr-Cl excimer lamp also emits UVC light having a wavelength of 230 nm or more. SafeZoneUVC® effectively eliminates UVC light with a wavelength of 230 nm or more by incorporating an appropriate optical filter inside the unit and also utilizing an opaque guide to ensure that light is not dispersed beyond the target area.

SUMMARY:
The threat of MRSA and multi-drug resistant pathogens have been growing in recent years. A new means of countering the infectious threat is required and one such modality is the use of UV light for disinfection. The aim of the study is to proof the efficacy of the 222nm UV light in disinfection on patients with sacral sores. This is a first in human proof-of-concept study

DETAILED DESCRIPTION:
Recent outbreaks of Ebola and MERS, and in the trend of growing threat of MRSA and multi-drug resistant pathogens, it is clear that a new means of countering the infectious threat is needed - even the US, EU, and Korean hospitals with the latest facilities has failed to stop the spread of these pathogens inside their wards.

This novel "Harmless UV Light," operating within the "Safe Zone Wave Length," will be a disruptive technology to counter the growing threats of infectious diseases, such as multi-drug-resistant bacteria and also viruses such as Ebola, MERS and new type Influenza. It will be a disruptive device in that it aims to be applied to fast, effective and labor-free disinfection of living environments, such as hospital wards, airports, and other public spaces to stop the spread of pathogens. This research is the first human clinical trial using this device that will spearhead the development of this technology, providing the key starting clinical data which would be the lead to development for a wider range of indications and markets. Successful proof of concept will lead to the next stage collaboration of larger scale clinical trials, and trials targeting wider range of indications and markets, at NUHS.

ELIGIBILITY:
Inclusion Criteria:

1. patients with pressure sore estimate at 2 cm X 2 cm or bigger
2. Patients with grade 2 or 3 sacral sores

Exclusion Criteria:

1. Patient who has pressure sore exposing bone
2. Patient who are beyond the age limits
3. Patient who is septic
4. Patient with obviously infected wound / pus in the wound
5. Patient who is pregnant.

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-01-23 (Actual)

PRIMARY OUTCOMES:
Bacterial colony forming unit counts | Up to 2 weeks for completion of 4 sessions of UV therapy
  bacterial colony-forming unit (cfu) counts for the pre and post UV therapy swabs

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2016-10-16): https://cdn.clinicaltrials.gov/large-docs/68/NCT03526068/Prot_000.pdf